CLINICAL TRIAL: NCT00661817
Title: Integrated Weight Loss Technologies for Weight and Blood Pressure Control in Urban Clinics
Brief Title: Evaluating a Blood Pressure Reduction and Weight Loss Program in a Low Income, Ethnically Diverse Population (The Be Fit, Be Well [BFBW] Study)
Acronym: BFBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Graham Colditz, Niess-Gain Professor in the School of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 448; U01HL087071 (NIH); U01HL087071-01 (NIH); RFA-HL-007
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Hypertension
Keywords: Exercise; Physical Fitness; Patient Compliance; Health Behavior
MeSH Terms: conditions — Obesity; Hypertension; Motor Activity; Patient Compliance; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants in this group will receive usual medical care and reading materials on weight loss.
  Interventions: Behavioral: Usual Care and Reading Materials
- 2 (Experimental): Participants in this group will take part in the lifestyle modification program.
  Interventions: Behavioral: Lifestyle Modification Program

INTERVENTIONS:
Behavioral: Lifestyle Modification Program — Participants will receive a behavior change "prescription" and skills training, offered via the Internet or through a combination of tailored print materials and an interactive voice response system, together with support strategies to enhance the intensity of the interpersonal and social-environmental support.
  Other Names: ES+SS (Environmental Support + Social Support)
  Arms: 2
Behavioral: Usual Care and Reading Materials — Participants in this group will receive usual medical care provided by their own primary care providers. They will also receive the NHLBI's "Aim for a Healthy Weight" brochure at the baseline study visit and again at the beginning of Year 2.
  Arms: 1

SUMMARY:
Obesity is a serious health problem that is a contributing factor for heart disease and high blood pressure. This study will evaluate a lifestyle modification program that aims to encourage weight loss and improve the health of people with high blood pressure from low income and minority communities.

DETAILED DESCRIPTION:
Obesity is a serious health problem in the United States, particularly among lower income and racial and ethnic minority populations. These populations have a high risk of developing heart disease and high blood pressure, and obesity is likely a contributing factor for both conditions. African-Americans, in particular, experience an earlier onset of high blood pressure and suffer more severe health consequences as a result, than do other racial and ethnic groups. This study will evaluate the effectiveness of a lifestyle modification program that will focus on reducing blood pressure levels and encouraging weight loss among patients at community health centers that serve a primarily low-income, ethnically diverse population. Researchers will also evaluate the cost effectiveness of the lifestyle modification program.

This 2-year study will enroll people who have high blood pressure. Participants will attend a baseline study visit to complete health questionnaires. They will then be randomly assigned to either receive usual care along with printed materials about maintaining a healthy weight or take part in the lifestyle modification program that incorporates health information technologies. Participants assigned to the program will visit the BFBW study Web site several times a week to review educational and motivational information. They may receive automated weekly phone calls that will prompt them to answer questions and assist them in setting goals for losing weight and managing their blood pressure. A study researcher will call participants every 6 weeks to discuss any problems and to invite participants to take part in optional walking groups or other group activities. Participants will attend group support sessions every other month and will wear a pedometer to track their walking habits. For all participants, study visits will occur at baseline and Months 6, 12, 18, and 24. All visits will include weight and blood pressure measurements, health questionnaires, and physician referrals if needed.

ELIGIBILITY:
Inclusion Criteria:

* High blood pressure that is being treated with medication
* BMI between 30 and 50 kg/m2
* Weighs no more than 400 lbs
* Willing to change diet, physical activity levels, and weight
* Willing to be assigned to either study group
* Patient of a participating community health center with a record of at least one medical visit in the 12 months before study entry
* Primary care provider approval is needed for people with the following conditions: diabetes mellitus, a prior cardiovascular event more than 6 months before study entry, known stable cardiovascular or peripheral vascular disease

Exclusion Criteria:

* Experienced a heart attack, stroke, or an atherosclerotic cardiovascular disease (ASCVD) procedure in the 6 months before study entry
* Serious medical condition that is likely to interfere with an accurate measurement of weight, for which weight loss is not medically advisable, or that would cause weight loss (e.g., end-stage renal disease [ESRD] and on dialysis; diagnosis or treatment for cancer in the 2 years before study entry, other than non-melanoma skin cancer)
* Prior or planned bariatric surgery
* Use of FDA-approved prescription weight loss medication, including off label drugs (e.g., topiramate, bupropion, byetta) or over-the-counter orlistat in the 6 months before study entry
* Long-term use (i.e., in the 6 months before study entry) of medications likely to cause weight gain or prevent weight loss (e.g., corticosteroids, lithium, olanzapine, risperidone, clozapine)
* Pregnant or breastfeeding in the 6 months before study entry
* Plans to become pregnant in the 2 years after study entry
* Plans to relocate from the area in the 2 years after study entry
* Another member of household is a study participant or study staff member
* Principal investigator decides that the individual is not suitable for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | Measured at Year 2

SECONDARY OUTCOMES:
Reduction in blood pressure | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Graham A. Colditz, MD, DrPH, Principal Investigator — Washington University School of Medicine; Gary G. Bennett, PhD, Principal Investigator — Dana Farber Cancer Institute/Harvard School of Public Health; Karen M. Emmons, PhD, Principal Investigator — Dana Farber Cancer Institute/Harvard School of Public Health
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ritzwoller DP, Glasgow RE, Sukhanova AY, Bennett GG, Warner ET, Greaney ML, Askew S, Goldman J, Emmons KM, Colditz GA; Be Fit Be Well study investigators. Economic analyses of the Be Fit Be Well program: a weight loss program for community health centers. J Gen Intern Med. 2013 Dec;28(12):1581-8. doi: 10.1007/s11606-013-2492-3. Epub 2013 Jun 4. PMID 23733374
- [Derived] Warner ET, Glasgow RE, Emmons KM, Bennett GG, Askew S, Rosner B, Colditz GA. Recruitment and retention of participants in a pragmatic randomized intervention trial at three community health clinics: results and lessons learned. BMC Public Health. 2013 Mar 6;13:192. doi: 10.1186/1471-2458-13-192. PMID 23496916
- [Derived] Bennett GG, Warner ET, Glasgow RE, Askew S, Goldman J, Ritzwoller DP, Emmons KM, Rosner BA, Colditz GA; Be Fit, Be Well Study Investigators. Obesity treatment for socioeconomically disadvantaged patients in primary care practice. Arch Intern Med. 2012 Apr 9;172(7):565-74. doi: 10.1001/archinternmed.2012.1. Epub 2012 Mar 12. PMID 22412073
- [Derived] Yeh HC, Clark JM, Emmons KE, Moore RH, Bennett GG, Warner ET, Sarwer DB, Jerome GJ, Miller ER, Volger S, Louis TA, Wells B, Wadden TA, Colditz GA, Appel LJ. Independent but coordinated trials: insights from the practice-based Opportunities for Weight Reduction Trials Collaborative Research Group. Clin Trials. 2010 Aug;7(4):322-32. doi: 10.1177/1740774510374213. Epub 2010 Jun 23. PMID 20573639